CLINICAL TRIAL: NCT01410760
Title: Perfusion Computed Tomography Pilot Study in the NCRN FOXFIRE Clinical Trial to Determine Blood Flow to Liver Metastases
Brief Title: PERfusion CT in the FOXFIRE Trial to Study Blood Flow to Liver Metastases
Acronym: PERFORM
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/H0505/95
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Imaging study; Perfusion Computerised Tomography
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Perfusion CT scan — Patients in this imaging substudy of the FOXFIRE clinical trial will undergo a perfusion CT prior to FOXFIRE protocol therapy( Ox/MDG chemo alone for 12 cycles in arm A or OX+MDG chemo for 12 cycles with Yttrium 90 SIRshpheres liver radioembolisaton in arm B cycle 2) on Day 1/2 cycle 2, Day 1/2 cycle 3 and Day 1/2 cycle 5 chemotherapy.

SUMMARY:
The PERFORM study is a pilot study investigating the feasibility and usefulness of performing a novel CT (Computed Tomography)scanning technique called Perfusion CT(CTP) as an addition to normal CT scanning in patients recruited to the FOXFIRE trial. All patients recruited to FOXFIRE at the Oxford Radcliffe Hospitals and University Hospitals of Leicester will be invited to take part. FOXFIRE is a national randomised controlled trial in which patients with unresectable liver tumours secondary to colorectal cancer will receive treatment with standard chemotherapy alone, or with chemotherapy in combination with an internal radiotherapy treatment which delivers radioactive particles(SIR-spheres) to the liver via its own blood supply (radioembolisation). In the FOXFIRE study a normal CT scan would usually be performed prior to the start of treatment and also three months after the commencement of treatment to assess the cancer's response to treatment, particularly whether the tumour has changed in size as a result of treatment. Perfusion CT gives the normal information on changes in tumour size but also assesses whether the blood flow to the cancer has changed, which may allow earlier identification of treatment success compared to normal CT scans. All patients consenting to participate in the PERFORM study will undergo four perfusion CT scans: one before the treatment starts, and one at the start of each of the second, third and fifth cycles of chemotherapy. The aim is to determine the feasibility of measuring tumour perfusion for data analysis using perfusion CT and to establish if the tumour perfusion pattern at baseline or shortly after the start of therapy can predict response to radioembolisation or chemotherapy. This research is funded by the National Institute for Health Research Biomedical Research Centre in Oxford and Oxfordshire Health Services Research Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent to participate in the FOXFIRE clinical trial and have not yet started chemotherapy treatment in the trial.
* Serum creatinine and calculated glomerular filtration rate are less than the upper limit of normal (ULN) in blood tests performed up to 29 days before entry into the FOXFIRE clinical trial.
* Liver metastasis 1.0 to4.0 cm in cranio-caudal diameter on imaging performed up to 29 days before entry into the FOXFIRE clinical trial

Exclusion Criteria:

* True allergy to intravenous iodinated CT contrast
* Active medical or psychological illness that would render the patient unsuitable for the additional imaging proposed in this pilot study, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate to this voluntary study and acquisition of sufficient data for perfusion analysis | 2 years

SECONDARY OUTCOMES:
Correlation between the tumour perfusion pattern on perfusion CT studies at baseline and shortly after the start of therapy and morphological response by RECIST criteria on CT scan 3 months post therapy in both arms of the FOXFIRE trial. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ricky A Sharma, MB BChir, Principal Investigator — University of Oxford
Locations (1):
- Oxford Radcliffe Hospitals NHS Trust, Oxford, United Kingdom